CLINICAL TRIAL: NCT05286138
Title: STUDY MULTICENRIC OBSERVATIONAL, NO-PROFIT FOR THE INCIDENCE AND CHARACTERISTICS OF MALIGNANT NEOPLASIES IN PATIENTS WITH HEMOGLOBINOPATHY FOLLOWED IN ITALY
Brief Title: STUDY INCIDENCE AND CHARACTERISTICS OF MALIGNANT NEOPLASIES IN PATIENTS WITH HEMOGLOBINOPATHY FOLLOWED IN ITALY
Acronym: Tum001
Status: Recruiting | Type: Observational
Sponsor: Società Italiana Talassemie ed Emoglobinopatie (Other)
Responsible Party: Sponsor
Other Study IDs: Tum001
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Malignacy, Hemoglobinopathie

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Trial aims to increase the information available on the relevance of tumor pathology in hemoglobinopathies, updating the data relating to hepatocarcinoma and investigating which other tumors are more frequent in patients with hemoglobinopathies. Still, in relation to tumor pathology, the study will evaluate any differences between the different types of hemoglobinopathy and will investigate the association between the appearance of neoplasms and risk factors such as age, sex, iron accumulation markers, history of bone marrow transplant, and others.

DETAILED DESCRIPTION:
By providing targeted screening strategies, these data may contribute to the early identification of tumor pathology in hemoglobinopathies, and, by contributing to the identification of risk factors, to its prevention. They will also be able to contribute to understanding which therapeutic approaches in the case of cancer are most appropriate in this category of subjects.

To be able to go even deeper into understanding the possible link that exists between tumors and hemoglobinopathy, a further data collection (substudy) has been prepared in which additional and more detailed information will be collected in order to evaluate which is the percentage of patients who develop tumors compared to all those with hemoglobinopathy.

The risk of developing tumors will also be assessed for each hemoglobinopathy (transfusion-dependent beta-thalassemia, transfusion independent beta-thalassemia, hemoglobin H disease, sickle cell disease, microdrepanocytosis)

ELIGIBILITY:
Inclusion Criteria:

* Transfusion-dependent or independent beta-thalassemia, hemoglobin H disease, sickle cell anemia and microdrepanocytosis
* Current or previous malignant tumor pathology
* Availability of medical history including the most relevant clinical and instrumental data before the onset of cancer

Exclusion Criteria:

* - Other haematological diseases other than hemoglobinopathies
* Absence of neoplastic events in the clinical history
* Non-availability of relevant clinical and instrumental data

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living or deceased adult or pediatric (male and female) patients with transfusion-dependent (TDT) or independent (NTDT) beta-thalassemia, hemoglobin H disease, sickle cell anemia and microdrepanocytosis who have developed tumor disease during life.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2052-02-28 (Estimated)

PRIMARY OUTCOMES:
outcome 1 | ENROLLMENT STUDY
  Evaluate the number of patients with hemoglobinopathy followed at Italian centers that have developed neoplastic events in the last decades
outcome 2 | enrollment study
  Evaluate which neoplasms are most associated with hemoglobinopathies
outcome 3 | enrollment study
  Identify any risk factors for the onset of neoplasms in patients with hemoglobinopathies.

SECONDARY OUTCOMES:
outcome 4 | enrollment study
  To highlight the differences between the various hemoglobinopathies as regards the development and characteristics of neoplastic events
outcome 5 | enrollment study
  Evaluate the possible association between neoplastic events and martial accumulation parameters in the different hemoglobinopathies
outcome 6 | enrollment study
  Evaluate the incidence and prevalence of neoplasms with respect to the total population of patients with hemoglobinopathies
outcome 7 | enrollment study
  Evaluate the impact of neoplasms as a cause of death in patients with hemoglobinopathies compared to other causes
outcome 8 | enrollment study
  To evaluate the incidence rate of neoplasms in the total population of patients affected by hemoglobinopathies and in the various forms of hemoglobinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: RAFFAELLA ORIGA, MD, Principal Investigator — Azienda Ospedaliero Universitaria di Cagliari
Locations (1):
- Azienda Ospedaliera Universitaria Di Cagliari, Cagliari, Italy